CLINICAL TRIAL: NCT00044070
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Effects of YM872 on Lesion Volume as Measured by Diffusion, Perfusion, and FLAIR Magnetic Resonance Imaging in Patients With Acute Ischemic Stroke
Brief Title: A Study to Evaluate the Effects of YM872 on Stroke Lesion Volume in Acute Stroke Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 872-CL-003
Record Dates: First submitted 2002-08-16; First posted 2002-08-20 (Estimated); Last update posted 2006-04-03 (Estimated); Status verified 2006-03

CONDITIONS: Cerebrovascular Accident
Keywords: ARTIST; Acute ischemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — YM 872

INTERVENTIONS:
Drug: YM872 (zonampanel)

SUMMARY:
This study will investigate the effects of a potential neuroprotectant compound, YM872, in the treatment of acute ischemic stroke. The study will determine if a 24-hour infusion of YM872, given within 6 hours of stroke onset, reduces the ischemic lesion volume as measured by MRI at 28 days after the infusion is given. The clinical effects of YM872 will also be determined by neurological function and disability scores at follow up visits through Day 90 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have suffered an acute ischemic stroke and can be evaluated and treatment initiated within 6 hours after the onset of symptoms (Onset is defined as the time that which the patient was last seen in a normal state, or bedtime for unwitnessed strokes occurring during the night).
* Patients who have a three dimensionally measurable lesion compatible with an acute ischemic stroke measured using MRI.
* Patients who have a National Institutes of Health Stroke Scale (NIHSS) score of at least 7 but not more than 23 and who are conscious.
* Patients who are able to provide written informed consent or have consent provided by a legally authorized representative.
* Patients who are at least 18 years of age.
* Other criteria as specified in the study protocol

Exclusion Criteria:

* Patients who have received alteplase (t-PA) for the current stroke episode. It is assumed that all patients who are eligible will receive treatment with t-PA.
* Patients who have disability and functional limitations prior to the current stroke episode (e.g. deficit resulting from a prior stroke).
* Patients who have brain hemorrhage.
* Patients who have stroke of the brainstem or cerebellum.
* Patients who cannot be evaluated using MRI due to the presence of a pacemaker, claustrophobia, need for sedation, etc.
* Patients who have renal (kidney) disease or insufficiency.
* Patients who have active epilepsy or convulsions during the current stroke episode.
* Patients who are IV drug users or are inebriated.
* Patients who have a history of drug-related anaphylaxis.
* Patients who have taken sedatives, anticonvulsants, or any medication with sedating effects in the 10 days prior study enrollment.
* Patients who have taken more than 1.3 g of aspirin per day in the 2 days prior to enrollment.
* Patients who have a known vitamin hypersensitivity.
* Other exclusion criteria as specified by the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12; Study Completion 2003-01

CONTACTS AND LOCATIONS:
Locations (89):
- United States (60):
  - University of South Alabama Stroke Center, Mobile, Alabama
  - Phoenix Neurology Associates (Good Samaritan Hospital), Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Providence St. Joseph's Medical Center, Burbank, California
  - Grossmont Hospital, La Mesa, California
  - UCLA Emergency Medical Center, Los Angeles, California
  - Good Samaritan Hospital, San Jose, California
  - Santa Monica UCLA Medical Center, Santa Monica, California
  - John Muir Medical Center, Walnut Creek, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Bethesda Memorial Hospital, Boynton Beach, Florida
  - Holmes Regional Medical Center, Melbourne, Florida
  - University of Miami (Jackson Memorial Hospital), Miami, Florida
  - Florida Neurovascular Institute, Tampa, Florida
  - DNA Research (Dekalb Medical Center), Decatur, Georgia
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Parkview Hospital, Fort Wayne, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Louisville Neuroscience Research Center, Louisville, Kentucky
  - Cullicchia Neurology Clinic, LLP, Marrero, Louisiana
  - Johns Hopkins Medical Institute, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - New England Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Field Neurosciences Institute (St. Mary's Hospital), Saginaw, Michigan
  - Advanced Neurology Specialists (Benefis Healthcare Hospital), Great Falls, Montana
  - St. Patrick's Hospital & Health Sciences Center, Missoula, Montana
  - Washoe Comprehensive Stroke Center, Reno, Nevada
  - JFK Medical Center, Edison, New Jersey
  - Neurology Group of Bergen County (Valley Hospital), Ridgewood, New Jersey
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - VA Medical Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Buffalo General Hospital, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - St. Luke's Hospital, New York, New York
  - Ellis Hospital, Schenectady, New York
  - Stony Brook Hospital, Stony Brook, New York
  - All-Trials Clinical Research, LLC (Rowan Regional Medical Center), Winston-Salem, North Carolina
  - Metrohealth Medical Center, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Medical College of Ohio, Toledo, Ohio
  - St. Elizabeth Health Center, Youngstown, Ohio
  - Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center Stroke Institute, Pittsburgh, Pennsylvania
  - Chattanooga Neurology Associates (Erlanger Hospital), Chattanooga, Tennessee
  - Chattanooga Neurology Associates (Memorial Hospital), Chattanooga, Tennessee
  - St. Thomas Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas (Houston Medical Center), Houston, Texas
  - Neurology Associates, Inc. (St. Mary's Hospital), Richmond, Virginia
  - Virginia Beach General Hospital, Virginia Beach, Virginia
  - Stevens Memorial Hospital, Edmonds, Washington
  - Providence St. Peter Hospital, Olympia, Washington
  - Sacred Heart Medical Center, Spokane, Washington
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Theda Clark Medical Center, Neenah, Wisconsin
- Universitätsklinik Allgemeines, Vienna, Austria
- Belgium (3):
  - Hopital Erasme, Brussels
  - Service de Neurologie, Cliniques Universitaires St.-Luc, Brussels
  - Dienst Neurologie UZ Gasthuisberg, Leuven
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Toronto Western Hospital, Toronto, Ontario
- Germany (13):
  - Universitätsklinikum Aachen, Neurologische Klinik, Aachen
  - Universität zu Köln klinik und poliklinik fur neurology, Cologne
  - University of Essen, Essen
  - Neurologische Universitätsklinik, Albert-Ludwigs-University, Freiburg im Breisgau
  - Universitätskrankenhaus Hamburg-Eppendorf Klinik für Neurologie, Hamburg-Eppendorf
  - Universitatklinikum Homburg, Neurologie Klinik und Poliklinik, Homburg Saar
  - Friedrich-Schiller-University, Jena
  - Universitatklinikum Leipzig, Leipzig
  - Universitätsklinik Mainz, Mainz
  - Department of Neurology Klinikum, Minden
  - Neurologische Klinik Klinikum Rechts der Isar der TU Munchen, München
  - Neurologische Klinik Knappschafts - krankenhause, Recklinghausen
  - Dr.-H.-Schmidt-Kliniken Ludwig-Erhar, Wiesbaden
- South Africa (9):
  - Muelmed Hospital, Arcadia
  - Bloemfontein Medi-Clinic, Bloemfontein
  - Groote Schuur Hospital, Cape Town
  - St. Augustine's Hospital, Durban
  - Sandton Medi-Clinic, Johannesburg
  - Pietermaritzburg Medi-Clinic, Pietermaritzburg
  - Little Company of Mary Medical Centre, Pretoria
  - Vergelegen Medi-Clinic, Somerset West
  - Sunninghill Hospital, Sunninghill